CLINICAL TRIAL: NCT02732314
Title: Efficacy and Tolerability of New Topical Formulations in Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Procter & Gamble Beauty (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSD2016003
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Dermatitis, Atopic; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Investigational OTC Cream (Experimental): Investigational OTC Cream applied topically, twice daily, for 12 weeks, once in the morning and once in the evening, to atopic dermatitis lesions and anywhere else the patient would apply their ordinary body moisturizer.
  Interventions: Drug: Investigational OTC Cream
- Placebo Cream (Placebo Comparator): Placebo Cream applied topically, twice daily, for 12 weeks, once in the morning and once in the evening, to atopic dermatitis lesions and anywhere else the patient would apply their ordinary body moisturizer.
  Interventions: Other: Placebo Cream
- Cosmetic Eczema Cream (Active Comparator): Cosmetic Eczema Cream applied topically, twice daily, for 12 weeks, once in the morning and once in the evening, to atopic dermatitis lesions and anywhere else the patient would apply their ordinary body moisturizer.
  Interventions: Other: Cosmetic Eczema Cream
- 0.05% Desonide Cream (Active Comparator): Rx Steroid applied topically, twice daily, once in the morning and once in the evening, for 4 weeks to atopic dermatitis lesions and then on any new lesions that appear for 4 weeks and as directed by the study doctor.
  Placebo Cream applied topically, twice daily, for 12 weeks, once in the morning and once in the evening, anywhere the patient would apply their ordinary body moisturizer except atopic dermatitis lesions.
  Interventions: Drug: 0.05% Desonide Cream; Other: Placebo Cream

INTERVENTIONS:
Drug: Investigational OTC Cream
  Arms: Investigational OTC Cream
Other: Cosmetic Eczema Cream
  Other Names: CeraVe
  Arms: Cosmetic Eczema Cream
Drug: 0.05% Desonide Cream
  Other Names: Actavis
  Arms: 0.05% Desonide Cream
Other: Placebo Cream
  Arms: 0.05% Desonide Cream; Placebo Cream

SUMMARY:
This is a 13 week randomized, double blind, parallel group, in home use study among approximately 60 male and female subjects, ages 12 to 65 years old inclusive, with atopic dermatitis (AD) SCORAD >16. Treatment group assignments will be balanced by disease severity, age, and body location of AD lesions. The study will consist of a 1 week washout phase and 12 week treatment phase. During the washout phase, subjects will be provided with a bar soap for bathing and showering and must refrain from using any other products on their body (excluding the face) including topical corticosteroids, ointments, lotions, sunscreens, etc. During the treatment phase, subjects will be randomized to 1 of 4 test legs. Throughout the treatment phase, the subjects will be required to use only the provided bar soap for bathing and showering and will apply their test product twice per day, once in the morning and once in the evening. No additional creams, moisturizers, lotions or cleansers other than those provided will be permitted for the duration of the study. Normal facial or hair care products are permitted, however, they must not contain anti-bacterial ingredients (e.g. antidandruff shampoo, acne products, etc).

SCORAD, EASI and PGA will incorporate whole body assessments. However, at the Baseline visit, subjects will have an active inflammatory lesion site and adjacent non-lesion, non-inflammatory site identified and marked for all instrumental and biopsy evaluations at Baseline and subsequent visits. Instrumental evaluations, imaging, expert visual grading and self-assessments will be performed throughout the study. Tolerability will be evaluated by incidence of AE's (defined per CTCAE), exacerbation of AD lesions, application site reactions/infections, and lab evaluations throughout the study. There will be additional consumption and compliance checks as well as dermatologic evaluations to ensure the subject's condition does not become extensively worse at each visit. A subset of subjects will have 2mm punch biopsies collected from the designated lesion and non-lesion sites at 3 time points throughout the study. The subset of subjects will be determined by subject willingness to participate in the biopsy portion as well as dermatologic evaluation and determination of biopsy candidacy.

ELIGIBILITY:
Inclusion Criteria:

* Is a generally healthy, male or female, 12-65 years old, inclusive
* Diagnosis of moderate or greater Atopic Dermatitis as determined by the Physician's Global Assessment (PGA of 3 or 4)

Exclusion Criteria:

* Is currently participating or has participated in another interventional clinical study at this or any other facility in the past 2 weeks
* Currently or has been diagnosed or treated for cancer in the past 5 years.
* Requires any topical or systemic medications that could affect the course of their atopic dermatitis during the study period (except inhaled steroids and/or stable antihistamines for asthma or allergies).
* Has a known hypersensitivity to any corticosteroid creams.
* Has a known sensitivity to Epinephrine, Xylocaine or topical antibiotics.
* Has a wound healing or blood-clotting abnormality.
* Has any active infections or has used antibiotics in the past 7 days.
* Has any physical attributes or skin conditions that might interfere with the clear visual or instrumental assessments.(i.e. cuts, sunburn, birth marks, tattoos, extensive scarring, excessive hair growth or acne)
* Has an immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS, lupus rheumatoid arthritis) which could place the subject at risk or interfere with the accuracy of the study results.
* Has used any immunosuppressant drugs or immunotherapy within the past 30 days or 5 half-lives.
* Is an employee of the Sponsor Company or clinical testing site.
* Is diabetic.
* Is dependent on oral medication for any skin disease/condition or could not, in the opinion of the Investigator tolerate the restriction of discontinuing the medicine as required in this study.
* Is currently pregnant or lactating or planning to become pregnant in the next 6 months.
* Has a history of keloid formation following skin injury.
* Is routinely taking anti-coagulant medications (i.e. Plavix, Coumadin, warfarin, heparin, etc.)
* Any other condition or factor the Investigator or their duly assigned representative believes may affect the ability of the subject to complete the study or the interpretation of the results.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
SCORAD (Severity Scoring of Atopic Dermatitis) | Change from Baseline at Week 12
  Dermatologic assessment and scoring of atopic dermatitis lesion severity

SECONDARY OUTCOMES:
SCORAD (Severity Scoring of Atopic Dermatitis) | Change from Baseline at Week 2
  Dermatologic assessment and scoring of atopic dermatitis lesion severity
SCORAD (Severity Scoring of Atopic Dermatitis) | Change from Baseline at Week 4
  Dermatologic assessment and scoring of atopic dermatitis lesion severity
SCORAD (Severity Scoring of Atopic Dermatitis) | Change from Baseline at Week 8
  Dermatologic assessment and scoring of atopic dermatitis lesion severity

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Nasir, MD, PhD, Principal Investigator — Wake Research Associates, LLC
Locations (1):
- Wake Research Associates, LLC, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No